CLINICAL TRIAL: NCT02419898
Title: Oxfordshire Women and Their Children's Health- A Feasibility Study
Brief Title: Oxfordshire Women and Their Children's Health
Acronym: OxWATCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Ingrid Granne, Senior Research Fellow in Reproductive Medicine, Oxford University Hospitals NHS Trust
Other Study IDs: 12/SC/0492
Record Dates: First submitted 2015-01-20; First posted 2015-04-17 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy; Pre-eclampsia; Gestational Diabetes; Depression; Metabolic Disorders; Pregnancy Induced Hypertension; Cardiovascular Disorders
Keywords: Feasibility
MeSH Terms: conditions — Pre-Eclampsia; Diabetes, Gestational; Depression; Metabolic Diseases; Hypertension, Pregnancy-Induced; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SST Serum, Citrate Platelet Free Plasma, EDTA Plasma, whole blood for DNA extraction, urine and saliva will be stored at -80°C for future studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Feasibility Study: Nulliparous women of reproductive age (18-40 years), who are not pregnant but could have a planned or unplanned pregnancy during the duration of the study.

SUMMARY:
The aim of this feasibility study is to test recruitment of participants into Phase 1 of the study and then the re-recruitment and retention of participants in Phase 2 of the study. The investigators will also be assessing the acceptability of recruitment strategy and data collection to participants.

The effect of pre-pregnancy factors (biophysical, genetic, socioeconomic, behavioural and psychological) on obstetric, cardiovascular, socioeconomic, behavioural and psychological outcomes will all be examined.

DETAILED DESCRIPTION:
The aim of this study is to recruit 300 women. The investigators anticipate that a subset of recruits will become pregnant during the pilot study.

This is a feasibility study with two phases:

* Phase 1: A detailed characterisation of nulliparous women who have an address in Oxfordshire or work in Oxfordshire
* Phase 2: Detailed assessment of events during and immediately after a first viable pregnancy.

During the Phase 1 visit:

* Participation is explained by a research nurse/midwife, any questions are answered and women, who agree, sign the consent form.
* A questionnaire covering medical and family history, socioeconomic information, behavioural factors and psychological measures will be completed.
* Baseline anthropometry - height, weight, hip/ waist ratio, USS measurement of fat (thigh and abdomen), bioimpedence.
* Cardiovascular - pulse and BP (peripheral / central), arterial stiffness, echocardiogram, carotid imaging and endothelial function (endo-check) tests are completed.
* Fasting venous blood sample (maximum 40 mls) including whole blood for maternal DNA.
* Urine sample
* Salivette

Once a participant has become pregnant she is eligible to enter phase 2 of the study. Phase 2 involves 6 further visits at 7, 11-13, 18-20, 28, 34 weeks gestation and 3 months post-delivery. During these visits repeated measurements of the above investigations will be carried out.

In addition, there will be a fetal ultrasound at 7 and 28 weeks and questionnaires at 7, 28 and 3 months post-delivery. An acceptability questionnaire will also be given to participants following completion of the study.

The end of the feasibility study will be the date of the final phase 2 visit of the last participant becoming pregnant during the feasibility study.

By collecting the above data the investigators anticipate recording and reporting longitudinal data in relation to the following:

•Incidence of obstetric complications

The incidence of pre-eclampsia, gestational diabetes, pregnancy induced hypertension, antenatal and postnatal depression and preterm birth.

•Longitudinal variation in cardiovascular parameters

Changes in longitudinal measures of blood pressure, carotid intima media thickness, pulse wave velocity, cardiac structure and function and endothelial function from pre-conception until 34 weeks gestation.

•Longitudinal changes in socioeconomic factors

By use of a questionnaire at pre-conception, 7 weeks gestation and 28 weeks gestation we will record employment and relationship status.

•Longitudinal changes in behavioural factors

By use of a questionnaire at pre-conception, 7 weeks gestation and 28 weeks gestation the investigators will record diet, weight control and perception, exercise, smoking, alcohol use and drug use.

•Longitudinal changes in psychological factors

By use of a questionnaire at pre-conception, 7 weeks gestation and 28 weeks gestation the investigators will record levels of anxiety, depression and quality of life and perceived health status.

•Longitudinal changes in the health status of participant and their family

By use of a questionnaire at pre-conception the investigators will record the participants' medical and family history, reproductive and sexual history and pain perception. At 7 weeks gestation and 28 weeks gestation the questionnaire will enquire about any changes or additions to the participants' medical and family history as well as reproductive and sexual health and pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant is female, aged 18-40 years
* Participant is not pregnant
* Participant lives or works in Oxfordshire

Exclusion Criteria:

* A previous live birth or still birth after 24 weeks gestation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be nulliparous women of reproductive age (18-40 years), who are not pregnant but could have a planned or unplanned pregnancy during the duration of the study. Participants must be willing to have research investigations before, during and after pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-04; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | 2 years
  This will be measured by the number of participants recruited into Phase 1 (pre-pregnancy) and Phase 2 (pregnancy) of the study. The investigators intend to recruit 300 participants into Phase 1 and 100 participants into Phase 2.

SECONDARY OUTCOMES:
The retention of participants in Phase 2 | 2 years
  The investigators aim to retain 90% of participants recruited into Phase 2 from 7 weeks gestation until delivery.
Incidence of pregnancy within 12 months of recruitment. | 2 years in total, 12 month for each recruit
Live birth rate | 2 years
Incidence of miscarriage and ectopic pregnancy in Phase 2 participants | 2 years
Incidence of loss to follow-up | 2 years
Proportion of participants who provide full data at baseline and throughout pregnancy | 2 years
Acceptability of the recruitment strategy to participants | 2 years
  At the end of a participant's involvement in the study the participant will be asked to complete an anonymous, validated acceptability questionnaire. It is anticipated that this will provide insight into why participants took part, the acceptability of the recruitment strategy, the participant's reactions to research participation and how acceptable the participant found study requirements and assessments.
Acceptability of the data collection procedures to participants. | 2 years
  At the end of a participant's involvement in the study the participant will be asked to complete an anonymous, validated acceptability questionnaire. It is anticipated that this will provide insight into why participants took part, the acceptability of the recruitment strategy, the participant's reactions to research participation and how acceptable the participant found study requirements and assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Granne, Principal Investigator — University of Oxford
Locations (1):
- The Nuffield Department of Obstetrics and Gynaecology, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harrison S, Petkovic G, Chevassut A, Brook L, Higgins N, Kenworthy Y, Selwood M, Snelgar T, Arnold L, Boardman H, Heneghan C, Leeson P, Redman C, Granne I. Oxfordshire Women and Their Children's Health (OxWATCH): protocol for a prospective cohort feasibility study. BMJ Open. 2015 Nov 9;5(11):e009282. doi: 10.1136/bmjopen-2015-009282. PMID 26553837